CLINICAL TRIAL: NCT00960167
Title: A Phase I Dose Escalation Trial of Conformal Hypofractionated Radiation Therapy for Patients With Hepatitis B Virus-Related Child A Cirrhosis and Hepatocellular Carcinoma
Brief Title: A Dose Escalation Trial of Radiation Therapy (RT) for Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Jason Chia-Hsien Cheng, Department of Oncology, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200906051R
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; radiotherapy; dose escalation; Toxicity; Local control
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiotherapy, Intensity-Modulated; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Level I (Experimental): 42 Gy in 12 fractions.
  Interventions: Radiation: 3DCRT or IMRT
- Dose Level II (Experimental): 49 Gy in 14 fractions.
  Interventions: Radiation: 3DCRT or IMRT
- Dose Level III (Experimental): 56 Gy in 16 fractions.
  Interventions: Radiation: 3DCRT or IMRT
- Dose Level IV (Experimental): 63 Gy in 18 fractions.
  Interventions: Radiation: 3DCRT or IMRT

INTERVENTIONS:
Radiation: 3DCRT or IMRT — All enrolled patients will receive 3.5 Gy per fraction (five fractions per week) at the following levels;
  Dose escalation by 7 Gy in 2 fractions to maximum of 63 Gy, as follows:
  Dose Level I: 3.5 Gy for 12 fractions (42 Gy total) Dose Level II: 3.5 Gy for 14 fractions (49 Gy total) Dose Level III: 3.5 Gy for 16 fractions (56 Gy total) Dose Level VI: 3.5 Gy for 18 fractions (63 Gy total)
  Other Names: Radiotherapy

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the leading malignancies in Taiwan. Surgery and local ablative therapy remain the treatment of choice for curative purpose. Transarterial chemoembolization has been the mainstay of intrahepatic control for patients not being candidates for local modalities of treatment. Sorafenib is recently integrated into the treatment options, mainly for intrahepatic or extrahepatic wide spread disease contraindicated for the other modalities. External radiotherapy (RT) has been selectively used for patients with the localized hepatic tumor(s) refractory to the above treatment options. The data from the retrospective studies were biased by the patient selection and uncontrolled comparison with patients not receiving RT. The obstacles for RT to HCC remain unanswered with heterogeneity in dose of radiation and lower tolerance of liver to RT in viral hepatitis carriers. Such a sublethal dose might be associated with unsatisfactory tumor control, intra-/extra-hepatic metastasis, and radiation-induced liver disease in a significant proportion of HCC patients.

The purposes of this phase I study are primarily to determine the maximally tolerated dose of RT, and secondarily to evaluate the tumor control, to assess patterns of failure and survival, to analyze the characteristics of radiation-induced liver disease, as well as to collect blood samples for translational research. HCC patients who are hepatitis B virus carriers and graded as Child-Pugh A cirrhosis are enrolled. This dose escalation trial is conducted with the 7-Gy increase in 2 fractions (3.5 Gy per fraction) for a total of four levels, from 42 Gy up to 63 Gy. Conformal RT with three-dimensional design, intensity modulated RT, or volumetric modulated arc therapy is used with the defined dose-volume threshold for normal liver and the other structures. Five patients are treated for each dose level, with dose limiting toxicity in less than 2 patients judged to be acceptable. A minimum of 15 patients are required for the starting dose level of 49 Gy if the treated tumor diameter is less than 10 cm. Imaging modalities are used for estimating treatment response and detecting metastasis. Serum analyses are done for evaluating hepatic function, viral load, hematological toxicity, and translational research for angiogenic and inflammatory studies.

DETAILED DESCRIPTION:
Synopsis

All enrolled patients will receive 3.5 Gy per fraction (five fractions per week) at the following levels;

Dose escalation by 7 Gy in 2 fractions to maximum of 63 Gy, as follows:

Dose Level I: 3.5 Gy for 12 fractions (42 Gy total) Dose Level II*: 3.5 Gy for 14 fractions (49 Gy total) Dose Level III: 3.5 Gy for 16 fractions (56 Gy total) Dose Level VI: 3.5 Gy for 18 fractions (63 Gy total) *Protocol treatment begins at level 2 for patients with the sum of the diameters of irradiated tumor(s) less than 10 cm.

Patient population:

Hepatocellular carcinoma based on the diagnostic criteria of European Association for the Study of the Liver (EASL), either confirmed cyto-histologically or confirmed non-invasively (restricted to cirrhotic patients) by radiological criteria (two coincident imaging techniques and focal lesion >2 cm with arterial hypervascularization) or combined criteria (one imaging technique associated with alpha-fetoprotein (AFP), focal lesion >2 cm with arterial hypervascularization, and AFP levels >400 ng/ml); Hepatitis B virus carrier serologically; Child-Pugh grade A for cirrhosis; The patients should be considered not suitable for surgery, ablation therapy, or trans-arterial chemoembolization judged by the caring physician. In addition, no systemic anti-cancer therapy with high priority is available judged by the caring physician.

Required sample size: Minimum of 15 (if starting from level II)

OBJECTS

Primary To identify the maximally tolerated dose (from 42 Gy up to 63 Gy in 3.5 Gy per fraction), conformal radiation therapy in patients with HBV-related Child-Pugh grade A cirrhosis and hepatocellular carcinoma (HCC) who are not eligible for other conventional treatment modalities.

Secondary To evaluate the local tumor control rate within the irradiated fields. To assess patterns of failure and survival of patients treated with conformal liver radiation therapy.

To analyze the dose volume characteristics that influence whether radiation-induced liver disease (RILD), HBV reactivation, or other toxicities occur.

To collect blood samples for translational research.

RADIATION THERAPY:

Radiation therapy must start within 4 weeks of patient registration. Intensity modulated radiation therapy or volumetric modulated arc therapy is acceptable. Helical tomotherapy or cyberknife is not allowed in this study. H2 blockers or proton pump inhibitors will be required in an attempt to reduce the risk of late gastrointestinal bleeding. Oral anti-viral agents are allowed at the discretion of the treating physician to prevent the reactivation of HBV.

Dose specification

The target dose is determined based on the study dose level and the volume of normal liver excluded from radiation, using the liver dose-volume histogram (DVH). Treatment at the allocated dose level is only permitted if the normal tissue criteria are maintained. If the normal tissue criteria are not met at that dose, treatment at a lower dose level is permitted, as long as the normal tissue constraints are met at the lower dose level.

The dose per fraction to the planning target volume (PTV) is 3.5 Gy. Dose will start at dose level 2 (49 Gy), but may vary from 42 Gy to 63 Gy, in 12 to 18 fractions, Monday through Friday, in 2-fraction increments. The starting level will be Level 2, 49 Gy in 14 fraction for patients with the sum of the diameters of irradiated tumor(s) less than 10 cm and Child-Pugh grade A of liver cirrhosis, and level 1, 42 Gy in 12 fraction for patients otherwise.

Doses will be prescribed to a peripheral covering isodose covering the PTV. Assuming dose is normalized to this isodose at 100%, the maximal dose can be 120% and the minimum PTV dose 90%. Any dose > 110% must be within the PTV (except for adjacent tumors, in which the maximum dose outside the PTV must be < 115%). Minor variation is defined as minimum PTV dose falling between 85 and 90% (of the required 100% isodose prescription). Major variation (unacceptable) is defined as minimum PTV dose < 85 % (for the required 100% isodose prescription). The acceptable exception is the underdose of PTV adjacent to small bowels to keep less than any 3cc of small bowels or stomach with the dose more than 42 Gy. This part of PTV should be specified and recorded.

Maximum doses are defined at 1 cc of volume. Minimum dose to the PTV is defined as minimum dose to 99.0% of the PTV.

*Protocol treatment begins at level 2 for patients with the sum of the diameters of irradiated tumor(s) less than 10 cm and Child-Pugh grade A of liver cirrhosis.

The minimum, maximum, and mean dose to the PTV is to be recorded for each gross tumor volume (GTV).

Technical factors

External beam equipment: Treatment will be delivered with 6 - 25 MV photons, with selection of appropriate energies to optimize the radiotherapy dose distribution within the target volume and minimize the dose to non-target tissues.

Localization, simulation and immobilization Patient positioning will be based on clinical judgment to best achieve the ideal dose distribution.

The target volume will be identified on an IV contrast CT scan and/or MRI that is registered to the planning CT dataset. The planning CT and all subsequent CT studies will be obtained using the identical immobilization technique used for treatment.

An immobilization frame may be used, but is not required. A variety of immobilization methods may be utilized for planning and treatment, including active breathing control (ABC), voluntary breath hold, gating, shallow breathing, or abdominal compression. For free breathing, 4D-CT can be used to aid in PTV definition.

Treatment planning/volume definitions

CT-based 3D treatment planning shall be used for all patients. Intensity modulated radiation therapy (IMRT) can be used for selected patients with breathing control device during IMRT.

The GTV will be defined by IV contrast CT or MRI. The clinical target volume (CTV) will be the GTV + 5 mm, within the liver. The PTV will be determined by the immobilization device used and/or the individual patient breathing motion. The minimal and maximal PTV margins permitted are 4 mm and 30 mm, respectively, dependent on the immobilization method used and breathing motion.

DVH shall be calculated for the liver (liver minus the GTVs), both kidneys, the spinal cord, small bowels and stomach as well as the target lesions (GTVs. CTVs, and PTVs). The maximum, minimum, and mean dose and dose per fraction must be documented.

Critical structures

Normal liver: The normal liver is defined as the normal liver volume minus GTV. In all patients, it is required that there is at least 700 cc of normal liver. No more than 30% of the normal liver may receive more than 27 Gy, and no more than 50% of normal liver may receive over 24 Gy.

Kidney: No more than 50% of the combined renal volume may receive 20 Gy or more.

Spinal cord: Maximal permitted dose to spinal cord is 37 Gy. Small bowel: Maximal permitted dose to small bowel is 42 Gy for any 3 cc volume. The underdose of PTV adjacent to small bowels or stomach is acceptable.

Stomach: Maximal permitted dose to stomach is 42 Gy for any 3 cc of volume. All doses are physical doses (not biologically corrected). Note that 42 Gy is biologically equivalent to 56.8 Gy in 2 Gy/fraction using an α/β of 3.

Radiation adverse events

Liver: Radiation therapy should be held at any point in the protocol for CTCAE v3.0 hepatic adverse event Grade 4. It is expected that a proportion of patients will have transient elevation of liver enzymes following treatment (possibly up to Grade 3 CTCAE levels). If elevation of liver enzymes is observed up to Grade 3 levels, more frequent measurements (at least once a week) of the liver enzymes are recommended until the enzymes stabilize or return to baseline levels. Repeat of all Grade 4 blood work is required at least 5 days following the first abnormal lab value to determine if the Grade 4 levels are transient (defined here as < 5 days) or persistent. Patients will be evaluated at 1-month and 3-month follow-up visits for symptoms and signs of radiation induced liver disease (RILD). In patients who have elevation of liver enzymes near Grade 4 levels and/or in patients with early non-specific signs or symptoms of liver injury, close follow-up is recommended with repeat blood work. If no tumor progression is documented in these patients, liver injury will be presumed to be treatment related.

HBV-related hepatitis: HBV-related hepatitis flare is defined as a greater than 3-fold increase of pre-treatment baseline serum ALT level and more than 100 IU/L. The HBV-related hepatitis flare (HBV reactivation) should be accompanied with the preceding or simultaneous greater than 10-fold increase, compared with previous nadir levels, of HBV DNA or by the reappearance of hepatitis B e antigen (HBeAg) in the serum of patients whose baseline HBeAg is negative. Oral anti-viral agent should be initiated in patients without prophylactic use of oral antiviral agents after HBV reactivation is confirmed.

Gastrointestinal: The dose constraints required for the normal stomach and small intestine should limit the GI toxicity observed and it is not expected that GI toxicity will be dose limiting. However, if a portion of the stomach or small intestine is treated (> 30 Gy), H2 blockers or proton pump inhibitors will be required to attempt to decrease the chance of late GI bleeding. Patients will be followed for GI toxicity at each follow up visit.

Other: The occurrence of Grade 4 adverse events, related to protocol treatment, in any organ system will prompt discontinuance of protocol therapy while appropriate physical examination, laboratory, and imaging assessments are undertaken. Protocol treatment will not be resumed in the absence of recovery from adverse events of this magnitude. Once recovery to grade 1 has occurred, treatment may continue at the discretion of the treating physician.

Evaluation of partial and complete response will be based on the 3-month follow-up CT scan. Only very gross increase in tumor size seen in less than that time will be scored as progressive disease. Response to radiation may continue up to 12 months follow-up and time of maximal response will be recorded.

Measurement of Response

Response will be evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. The sum of the longest diameter (LD) for all target lesions will be calculated and reported as the baseline sum LD. The baseline sum LD will be used as reference by which to characterize the objective tumor.

Response Criteria: Evaluation of target lesions Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.

Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.

Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study

In-field local control: For this study, local control is defined as the lack of progressive disease in the treated fields.

Cause of death: The treating physician will evaluate whether the cause of death was hepatic or non-hepatic, and/or due to tumor or due to toxicity

SPECIMEN COLLECTION FOR TRANSLATIONAL RESEARCH

Peripheral Blood Collection

Sample collection time points:

Blood samples will be collected in 5 occasions along the protocol treatment:

1. baseline (within 1 week before the first radiotherapy fraction);
2. 5-10 days after the last radiotherapy fraction;
3. 4 weeks after the last radiotherapy fraction.

Preparation of Plasma and Buffy coat:

1. Collect 5-10 mL of anticoagulated blood (EDTA). Invert tube several times to assure blood is mixed thoroughly with anticoagulant.
2. Using three (3) 1mL cryovials, label them patient's case number, procedure date, and clearly mark cryovials "plasma". Similarly, label three (3) 1mL cryovials and mark as "buffy coat".

Process:

1. Centrifuge specimens within one hour of collection. EDTA (purple top) tubes should be centrifuged in a standard clinical centrifuge at ~2500 RPM at 4° Celsius for 10 minutes.
2. If the interval between specimen collection and processing is anticipated to be greater than one hour, keep specimen on ice until centrifuging is done.
3. Remove plasma close to the buffy coat taking cared not to disturb the white cell layer. Aliquot plasma into three 1mL cryovials labeled with the RTOG study and case numbers, procedure date, and clearly mark as "plasma".
4. Remove the buffy coat cells carefully and place into the 1 mL cryovials labeled "buffy coat" (it is okay if a few packed red cells below the buffy coat layer are inadvertently collected in the process)
5. Place cryovials into biohazard bag.
6. Store plasma and buffy coat specimens frozen. Buffy coat samples must be shipped to the tissue bank within one (1) week of collection.

Preparation of Serum:

1. Collect one 5-10 mL red-topped tube. Allow 30 minutes for clotting at room temperature before processing.
2. Using four (4) 1ml cryovials, label them with the study number, and patient's case number, procedure date, and clearly mark cryovials as "serum".

Process:

1. Allow one 5ml red top tube to clot for 30 minutes at room temperature.
2. Spin red-topped tube in a standard clinical centrifuge at ~2500 RPM at 4°Celsius for 10 minutes.
3. Aliquot serum into the four 1mL cryovials labeled with the RTOG study and case numbers, procedure date, and marked "serum".
4. Store serum frozen (at -80° Celsius) until ready to ship

Analysis of Blood Samples

Serum or plasma samples:

Soluble cytokines and growth factors related to inflammation and angiogenesis will be analyzed by enzyme-linked immunosorbent assay (ELISA) for serum samples and plasma samples. Inflammatory factors, such as IL-6, TNF-alpha, CRP, MMP-2, MMP-9, VEGF, IL-8, pro-angiogenic factors, such as VEGF, basic-FGF, PDGF, PIGF, and TNF, and anti-angiogenic factors, such as thrombospontin-1 (TSP-1), will be included. Serum HBV DNA level will also be analyzed.

RNA samples from blood mononuclear cells:

1. Tumor-associated gene expression in peripheral blood reflects the presence of circulating hepatocellular carcinoma (HCC) cells and might be associated with aggressive features of HCC. We will assess the prognostic significance of AFP and human telomerase reverse transcriptase protein (hTERT) mRNA expression in the peripheral blood of HCC patients.
2. Circulating endothelial cells and their progenitors have been shown as surrogate markers of angiogenic activity. Several cellular markers, including VEGFR2, Tie-2, and CD133, have been shown to be specifically expressed in activated endothelial cells or endothelial progenitor cells. The expression of these markers will be detected by real-time quantitative PCR.

DNA samples from blood mononuclear cells:

The polymorphic inheritance of human drug-metabolizing enzymes, such as those encoded by the glutathione-S-transferase (GST), microsomal epoxide hydrolase (mEPHX), and CYP systems, have been implicated in both cancer risk and prognosis. DNA samples from blood mononuclear cells will be used for the analysis of GST, mEPHX, CYP, and p53 polymorphism by PCR and sequencing analysis.

Data Management and Analysis

1. Evaluation of soluble factors related to inflammation or angiogenesis and the surrogate quantification of circulating endothelial cells or progenitors (the B-2 section) will be conducted according to standard procedures by personnel who have no access to the clinical outcomes of the patients.
2. The clinical outcomes of the patients will be included for further correlation study include clinical responses (responders vs. non-responders), other patterns of failure (intrahepatic recurrence outside radiation field vs. no intrahepatic recurrence; extrahepatic metastasis vs. no metastasis), radiation induced liver disease (RILD vs. no RILD), and survival.
3. The correlation of clinical outcomes with the surrogate markers evaluated from the after-mentioned markers will be made.

STATISTICAL CONSIDERATIONS

Study Endpoints The primary endpoint of this study is to determine the maximally tolerated dose of highly conformal radiation therapy in patients with HCC. The secondary endpoints are to evaluate local control rate within the irradiated fields,to assess patterns of failure and survival, and to analyze the dose volume characteristics that influence whether RILD, HBV reactivation, or other toxicities occur.

Sample Size

Evaluation of Adverse Events

Adverse events will be graded according to the CTCAE v. 3.0 criteria. Dose limiting toxicity (DLT) is defined as any of the following occurring within 90 days from the start of treatment:

a) grade 4 or 5 hepatic b) grade 4 or 5 gastrointestinal c) grade 4 or 5 thrombocytopenia d) Radiation Induced Liver Disease (RILD) requiring treatment (including diuretics). RILD will be defined using the following adverse events: i) grade 3 or higher alkaline phosphatase (ALP) in the presence of ascites occurring in the absence of disease progression ii) grade 4 hepatic liver enzyme elevations persisting for ≥ 5 days e) any adverse event requiring interruption of therapy by ≥ 2 weeks (14 calendar days). This does not include patient desire to discontinue therapy. It does include failure for thrombocytopenia to improve to a level of 80 requiring interruption of therapy.

f) Any grade 5 adverse event The goal of this study is to determine the maximally tolerated dose (MTD) for patients with HCC, such that the rate of DLT is less than 35%.

Dose Escalation

The following are the four possible dose levels for this study:

Dose Level I: 3.5 Gy for 12 fractions (42 Gy total) Dose Level II: 3.5 Gy for 14 fractions (49 Gy total) Dose Level III: 3.5 Gy for 16 fractions (56 Gy total) Dose Level VI: 3.5 Gy for 18 fractions (63 Gy total)

Patients will receive highly conformal radiotherapy starting at Dose Level II. Dose levels will be escalated by 7 Gy in 2 fractions per level up to 21 Gy in 6 fractions and a total dose of 63 Gy. Evaluable patients will be defined as any eligible patient that begins treatment. After 5 evaluable patients have been followed for a minimum of 90 days from the start of treatment, if there are 0 or 1 DLT, the dose level will be judged to be acceptable. If this occurs, then patients will begin to be accrued at the next higher dose level. If ≥ 3 of 5 patients have DLT, the preceding dose level will be declared to be the MTD. If 2 of 5 patients have DLT, the addition of 5 more patients to the same level will be done. If ≥ 4 of 10 patients have DLT, the preceding dose level will be declared to be the MTD. If 2 or 3 of the 10 patients have DLT, patients will begin to be accrued at the next higher dose level. If there are 3 or more DLT at the starting dose level (Dose Level II), then the dose will be de-escalated to Dose Level I. If this occurs, then after 5 evaluable patients have been followed for a minimum of 90 days from the start of treatment at Dose Level I, if there are 0 or 1 DLT, the 3.5 Gy per fraction for a total of 42 Gy will be declared to be the MTD. If at any time a grade 5 treatment-related adverse event is observed, the study chairs will review the event.

The number of evaluable patients that will be needed depends on the number of times the dose is escalated or possibly de-escalated. If the escalation continues up through Dose Level IV, 15 evaluable patients will be required. If the dose is de-escalated after Dose Level II, then 10 evaluable patients will be required.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients include those with HCC based on the diagnostic criteria of European Association for the Study of the Liver (EASL), either confirmed cyto-histologically or confirmed non-invasively (restricted to cirrhotic patients) by radiological criteria (two coincident imaging techniques and focal lesion > 2 cm with arterial hypervascularization) or combined criteria (one imaging technique associated with AFP, focal lesion > 2 cm with arterial hypervascularization, and AFP levels > 400 ng/ml).
* They have Child-Pugh grade A cirrhosis and are HBsAg-positive for more than 6 months.
* These patients are not feasible for other conventional treatment modalities of treatment including surgery, transarterial embolization, ethanol injection, and radiofrequency ablation.
* No systemic anti-cancer therapy with high priority is available.
* All of the above 3 criteria should be judged by the caring physician.
* All intrahepatic disease must be encompassed within the radiation fields, except intrahepatic diseases outside the radiation field(s) have been controlled by other treatment modalities before radiotherapy.
* Karnofsky Performance Scale ≧ 80.
* Age > 18.
* Adequate bone marrow function, defined as follows:

  * Absolute neutrophil count (ANC) > 1,000 cells/mm3 based upon CBC/differential obtained within 2 weeks prior to registration on study
  * Platelets > 20,000 cells/mm3 based upon CBC/differential obtained within 2 weeks prior to registration on study
  * Hemoglobin > 8.0 g/dl based upon CBC/differential obtained within 2 weeks prior to registration on study (Note: The use of blood transfusion or other intervention to achieve Hgb > 8.0 g/dl is acceptable.)
* Previous liver resection, embolization, or ablative therapy is permitted.
* Chemotherapy and/or targeted agent therapy must be completed at least 2 weeks prior to radiation.
* Women of childbearing potential and male participants must practice adequate contraception.
* Patient must sign informed consent prior to study entry.
* Pretreatment evaluations for eligibility include:

  * A complete history and general physical examination
  * For women of childbearing potential, a serum or urine pregnancy test must be performed within 72 hours prior to registration INR, total bilirubin, albumin, alkaline phosphatase, AST, ALT within 1 week prior to study entry
  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR at least 10 mm by spiral CT scan

Exclusion Criteria:

* Prior invasive malignancy, other than HCC, (except nonmelanomatous skin cancer) unless disease free for a minimum of 3 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
* Tumor thrombosis in the main trunk of portal vein, hepatic vein, or inferior vena cava.
* Child-Pugh grade B or C cirrhosis.
* Extrahepatic metastasis.
* Clinical ascites that requires diuretic treatment or paracentesis for symptom relief.
* Serum alanine aminotransferase (ALT) level > 5X normal upper limits or total bilirubin level > 3.0.
* Active hepatitis (serum ALT level > 5X normal upper limits) or clinically significant liver failure.
* Positivity of anti-HCV, pregnancy, nursing women, or women of childbearing potential, and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Maximally tolerated dose of RT | weekly during radiotherapy

SECONDARY OUTCOMES:
Tumor control, patterns of failure and survival | Monthly after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chia-Hsien Cheng, Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan